CLINICAL TRIAL: NCT01619930
Title: The Effects on Depression of Internet-administered Behavioural Activation and Physical Exercise With Treatment Rationale and Relapse Prevention: Study Protocol for a Randomised Controlled Trial
Brief Title: The Effects of Behavioral Activation and Physical Exercise on Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTUA
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Depression
Keywords: Depression; Behavioral activation
MeSH Terms: conditions — Depression | interventions — Exercise; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1a (Experimental): In phase 1, group 1 undergoes physical activation without added motivation interviewing. Post-treatment (phase 2), group 1 is divided by randomization into group 1a and 1b, where 1a receives relapse prevention and 1b does not. Both 1a and 1b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 1 + 12 from waiting list control group)
  Interventions: Behavioral: Physical activity without motivational interviewing
- 1b (Experimental): In phase 1, group 1 undergoes physical activation without added motivation interviewing. Post-treatment (phase 2), group 1 is divided by randomization into group 1a and 1b, where 1a receives relapse prevention and 1b does not. Both 1a and 1b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 1 + 12 from waiting list control group)
  Interventions: Behavioral: Physical activity without motivational interviewing
- 2a (Experimental): In phase 1, group 2 undergoes physical activation with added motivation interviewing. Post-treatment (phase 2), group 2 is divided by randomization into group 2a and 2b, where 2a receives relapse prevention and 2b does not. Both 2a and 2b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 2 + 12 from waiting list control group)
  Interventions: Behavioral: Physical exercise with motivational interviewing
- 2b (Experimental): In phase 1, group 2 undergoes physical activation with added motivation interviewing. Post-treatment (phase 2), group 2 is divided by randomization into group 2a and 2b, where 2a receives relapse prevention and 2b does not. Both 2a and 2b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 2 + 12 from waiting list control group)
  Interventions: Behavioral: Physical exercise with motivational interviewing
- 3a (Experimental): In phase 1, group 3 undergoes behavioral activation with added motivation interviewing. Post-treatment (phase 2), group 3 is divided by randomization into group 3a and 3b, where 3a receives relapse prevention and 3b does not. Both 3a and 3b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 3 + 12 from waiting list control group)
  Interventions: Behavioral: Behavioral activation with rationale
- 3b (Experimental): In phase 1, group 3 undergoes behavioral activation with added motivation interviewing. Post-treatment (phase 2), group 3 is divided by randomization into group 3a and 3b, where 3a receives relapse prevention and 3b does not. Both 3a and 3b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 3 + 12 from waiting list control group)
  Interventions: Behavioral: Behavioral activation with rationale
- 4a (Experimental): In phase 1, group 4 undergoes behavioral activation without added motivation interviewing. Post-treatment (phase 2), group 4 is divided by randomization into group 4a and 4b, where 4a receives relapse prevention and 4b does not. Both 4a and 4b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 4 + 12 from waiting list control group)
  Interventions: Behavioral: Behavioral activation without rationale
- 4b (Experimental): In phase 1, group 4 undergoes behavioral activation with added motivation interviewing. Post-treatment (phase 2), group 4 is divided by randomization into group 4a and 4b, where 4a receives relapse prevention and 4b does not. Both 4a and 4b undergo post-treatment measurements as previously described.
  n = 50 + 12 = 62 (50 from group 4 + 12 from waiting list control group)
  Interventions: Behavioral: Behavioral activation without rationale
- Phase 1 Waiting list control group (No Intervention): Control group during phase 1, in parallel with treatment groups 1-4. Weekly self-report measurements, the results of which are conveyed in the form of individualized feedback. After 12 weeks, the participants of the control group (n = 100) are randomized to one four phase 1 active treatment groups (1-4) and receive treatment accordingly.

INTERVENTIONS:
Behavioral: Physical activity without motivational interviewing — Focus is on physical exercise, motivated by research findings that it has a positive effect on depressive symptoms. An individualized exercise program is constructed, to be followed by the respective participant. A user-friendly pulse watch will be mailed to participants. Exercise is monitored through online self-registration with automated feedback.
  Arms: 1a; 1b
Behavioral: Physical exercise with motivational interviewing — Focus is on physical exercise, motivated by research findings that it has a positive effect on depressive symptoms. An individualized exercise program is constructed, to be followed by the respective participant. A user-friendly pulse watch will be mailed to participants. Exercise is monitored through online self-registration with automated feedback. An initial motivational interview (MI) per telephone is also conducted, to explore the intrinsic motivation to change in participants.
  Arms: 2a; 2b
Behavioral: Behavioral activation with rationale — A behavioral activation program, based on the TRAP-TRAC model according to which suffering individuals are trapped in a vicious circle of avoidance and ever fewer reinforcers, leading to increasing discomfort. To break free of this vicious circle, patients have to replace avoidance patterns with alternative coping strategies. Unlike previous applications of this program done in the U.S., this study will feature an internet-based administration. Approximately 15 minutes of electronic therapist support will be included per week.
  Arms: 3a; 3b
Behavioral: Behavioral activation without rationale — A behavioral activation program without TRAP-TRAC rationale, but with some encouragement provided ("Activate yourself and feel better!"). Approximately 15 minutes of electronic therapist support will be included per week.
  Arms: 4a; 4b

SUMMARY:
The purpose of this study is to compare an internet-based behavioral activation program with a physical activation program, as treatments for mild to moderate depression. The added effect of rationale and motivational interviewing will also be studied, as well as the effects of relapse prevention program.

DETAILED DESCRIPTION:
BACKGROUND:

Despite their potential as low-threshold, low-cost and high-flexibility treatments of depression, behavioural activation and physical exercise have not yet been directly compared. This study will examine the effects of these interventions, administered via the Internet. The added effect of providing a treatment rationale will also be studied, as well as a relapse prevention program featuring cognitive behavioural therapy components.

METHODS/DESIGN:

This randomised controlled trial will include 500 participants meeting the diagnostic criteria for major depression, recruited in multiple cycles and randomised to either a waiting list control group with delayed treatment, or one of the four treatment groups: (1) physical exercise without a clear treatment rationale; (2) physical exercise with treatment rationale; (3) behavioural activation with treatment rationale; or (4) behavioural activation without a clear treatment rationale. Post treatment, half of the participants will be offered a relapse prevention program. Primary outcome measure will be the Patient Health Questionnaire 9-item. Secondary measures include diagnostic criteria for depression, as well as self-reported anxiety, physical activity and quality of life. Measurements - done via telephone and the Internet - will be collected pre-treatment, weekly during treatment period, immediately post treatment and then monthly during a 24-month follow-up period.

DISCUSSION:

The results of this study will constitute an important contribution to the body of knowledge of the respective interventions.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV (or DSM-V) criteria for depression, with depression being primary diagnosis
* Scoring within the interval 15-35 on the Montgomery-Åsberg Depression Rating Scale (MADRS)
* Living in Sweden and being able to read Swedish
* Access to computer with internet connection

Exclusion Criteria:

* Currently receiving other psychological treatment
* Non-stable use of psychoactive medication
* Deemed to suffer from a too severe depression
* Deemed to suffer from other psychological disorder, e.g. psychosis, bipolarity etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Patient Health Questionnaire (PHQ-9) | Weekly during treatment period of 12 weeks
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 24 hours
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 12 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 24 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | Monthly, 0-24 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).

SECONDARY OUTCOMES:
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 24 hours
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 12 months
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 24 months
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | Monthly, 0-24 months
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | 24 hours
  The International Physical Activity Questionnaire is a measure of physical activity.
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | 12 months
  The International Physical Activity Questionnaire is a measure of physical activity.
Change from baseline in the International Physical Activity Questionnaire (IPAQ) | 24 months
  The International Physical Activity Questionnaire is a measure of physical activity.
Change from baseline in Quality Of Life Inventory (QOLI) | 24 hours
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 12 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 24 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in MINI | Monthly, 0-24 months
  The Mini International Neuropsychiatric Interview is a short, structured interview designed for clinicians to diagnose axel I DSM-IV and ICD-10 disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Department of Psychology, Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] Carlbring P, Lindner P, Martell C, Hassmen P, Forsberg L, Strom L, Andersson G. The effects on depression of Internet-administered behavioural activation and physical exercise with treatment rationale and relapse prevention: study protocol for a randomised controlled trial. Trials. 2013 Feb 2;14:35. doi: 10.1186/1745-6215-14-35. PMID 23374879
- [Derived] Hlynsson JI, Kristjansson T, Andersson G, Carlbring P; ACTUA research group. Evaluating the necessity of booster sessions in relapse prevention for depression: a longitudinal study. Front Psychol. 2025 Jun 24;16:1568141. doi: 10.3389/fpsyg.2025.1568141. eCollection 2025. PMID 40631058